CLINICAL TRIAL: NCT02864940
Title: MASH Study (Memory Training in Aneurysmal Subarachnoid Hemorrhage Patients)
Brief Title: Memory Training in Aneurysmal Subarachnoid Hemorrhage Patients
Acronym: MASH
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to enroll
Sponsor: Rush University Medical Center (Other)
Collaborators: Lumos Labs, Inc. (Industry)
Responsible Party: Principal Investigator, Michael Chen, M.D., Associate Professor of Neurology, Neurosurgery and Radiology, Rush University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MASH 14080402
Record Dates: First submitted 2016-08-05; First posted 2016-08-12 (Estimated); Results first posted 2023-04-10 (Actual); Last update posted 2023-04-10 (Actual); Status verified 2023-03

CONDITIONS: Ruptured Aneurysm; Memory Deficits; Subarachnoid Hemorrhage
Keywords: Memory; aneurysm; deficits; trouble; forgetful; ruptured; subarachnoid; hemorrhage
MeSH Terms: conditions — Aneurysm, Ruptured; Memory Disorders; Subarachnoid Hemorrhage; Aneurysm; Rupture; Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention Arm (Experimental): Using the cognitive exercises on Lumosity for 10 weeks
  Interventions: Device: Lumosity
- Control Arm (Active Comparator): Using online crossword puzzles for 10 weeks.
  Interventions: Device: Crossword puzzle

INTERVENTIONS:
Device: Lumosity — A web-based cognitive training platform that includes games designed with the purpose of improving the user's cognitive abilities
  Arms: Intervention Arm
Device: Crossword puzzle — This game offers a choice between three puzzle sizes, three levels of complexity, and varying font sizes. It also includes optional help features such as filling in an unknown letter or word.
  Arms: Control Arm

SUMMARY:
The study aim is to determine if periodic online cognitive exercises (Lumosity) improve memory function in ruptured cerebral aneurysm patients with disabling baseline memory deficits within the first 24 months after rupture. Half of the subjects will be randomized to use Lumosity-designed online cognitive exercises and half will serve as an active control group performing online crossword puzzles.

DETAILED DESCRIPTION:
In this prospective randomized, control clinical trial subjects have a self-reported disabling memory deficit within the first two years of their ruptured cerebral aneurysm. Subjects will be recruited in the neurosurgery clinic setting, via email and phone screen, through social media and phone screen, or during a monthly support group for the patient population in question.

During the screening interview the inclusion and exclusion criteria are assessed and informed consent is obtained if needed.

Those who qualify for the study will undergo a baseline assessment involving Checklist for cognitive and emotional consequences following stroke (CLCE-24), Working memory questionnaire, Activity of Daily living Questionnaire, and a Lumosity Administered assessment.

After baseline assessments randomization will occur stratified according to duration since SAH <12 or >12 months, to either a treatment group, which will include online access to structure-oriented activities (Lumosity), or an active control group(online crossword puzzles).

Subjects in the intervention group will undergo twenty training sessions over 10 weeks involving cognitive games selected from Lumocity. Games will be customized using an automated algorithm supplied by Lumosity, to determine performance in the various targeted skills, which include: task switching, logical reasoning, quantitative reasoning, response inhibition, numerical calculation, working memory, face-name recall, selective attention, spatial recall, spatial orientations, planning, and divided attention. The recommended duration of interaction is 2 hours per week for 10 weeks.

The control group uses a computerized crossword puzzle. the puzzle is offered in three different puzzle sizes, levels of complexity, and font sizes. these puzzles do not provide progressive challenge to the user by either increased speed, visual field size, number of distractors, or degree of difficulty of target stimulus differentiation.

ELIGIBILITY:
Inclusion Criteria:

* Ruptured cerebral aneurysm-confirmed by study personnel within past year
* Age 18 and older
* Those with a modified Rankin 0 or 1
* Baseline memory problem affecting daily life
* Home computer or tablet with internet access

Exclusion Criteria:

* Unable to read or speak English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2016-06; Primary Completion 2018-08-15 (Actual); Study Completion 2018-08-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brisman JL, Song JK, Newell DW. Cerebral aneurysms. N Engl J Med. 2006 Aug 31;355(9):928-39. doi: 10.1056/NEJMra052760. No abstract available. PMID 16943405
- [Background] Rinkel GJ, Algra A. Long-term outcomes of patients with aneurysmal subarachnoid haemorrhage. Lancet Neurol. 2011 Apr;10(4):349-56. doi: 10.1016/S1474-4422(11)70017-5. PMID 21435599
- [Background] Passier PE, Visser-Meily JM, van Zandvoort MJ, Post MW, Rinkel GJ, van Heugten C. Prevalence and determinants of cognitive complaints after aneurysmal subarachnoid hemorrhage. Cerebrovasc Dis. 2010;29(6):557-63. doi: 10.1159/000306642. Epub 2010 Apr 8. PMID 20375498
- [Background] Sheldon S, Macdonald RL, Schweizer TA. Free recall memory performance after aneurysmal subarachnoid hemorrhage. J Int Neuropsychol Soc. 2012 Mar;18(2):334-42. doi: 10.1017/S1355617711001780. Epub 2012 Feb 13. PMID 22325677
- [Background] Sheldon S, Macdonald RL, Cusimano M, Spears J, Schweizer TA. Long-term consequences of subarachnoid hemorrhage: examining working memory. J Neurol Sci. 2013 Sep 15;332(1-2):145-7. doi: 10.1016/j.jns.2013.06.021. Epub 2013 Jul 18. PMID 23871092
- [Background] Al-Khindi T, Macdonald RL, Schweizer TA. Decision-making deficits persist after aneurysmal subarachnoid hemorrhage. Neuropsychology. 2014 Jan;28(1):68-74. doi: 10.1037/neu0000003. Epub 2013 Sep 16. PMID 24040927
- [Background] Chen M, Mangubat E, Ouyang B. Patient-reported outcome measures for patients with cerebral aneurysms acquired via social media: data from a large nationwide sample. J Neurointerv Surg. 2016 Jan;8(1):42-6. doi: 10.1136/neurintsurg-2014-011492. Epub 2014 Dec 1. PMID 25452396
- [Background] Levine B, Schweizer TA, O'Connor C, Turner G, Gillingham S, Stuss DT, Manly T, Robertson IH. Rehabilitation of executive functioning in patients with frontal lobe brain damage with goal management training. Front Hum Neurosci. 2011 Feb 17;5:9. doi: 10.3389/fnhum.2011.00009. eCollection 2011. PMID 21369362
- [Background] Westerberg H, Jacobaeus H, Hirvikoski T, Clevberger P, Ostensson ML, Bartfai A, Klingberg T. Computerized working memory training after stroke--a pilot study. Brain Inj. 2007 Jan;21(1):21-9. doi: 10.1080/02699050601148726. PMID 17364516
- [Background] Willis SL, Tennstedt SL, Marsiske M, Ball K, Elias J, Koepke KM, Morris JN, Rebok GW, Unverzagt FW, Stoddard AM, Wright E; ACTIVE Study Group. Long-term effects of cognitive training on everyday functional outcomes in older adults. JAMA. 2006 Dec 20;296(23):2805-14. doi: 10.1001/jama.296.23.2805. PMID 17179457
- [Background] Ball K, Berch DB, Helmers KF, Jobe JB, Leveck MD, Marsiske M, Morris JN, Rebok GW, Smith DM, Tennstedt SL, Unverzagt FW, Willis SL; Advanced Cognitive Training for Independent and Vital Elderly Study Group. Effects of cognitive training interventions with older adults: a randomized controlled trial. JAMA. 2002 Nov 13;288(18):2271-81. doi: 10.1001/jama.288.18.2271. PMID 12425704
- [Background] Jobe JB, Smith DM, Ball K, Tennstedt SL, Marsiske M, Willis SL, Rebok GW, Morris JN, Helmers KF, Leveck MD, Kleinman K. ACTIVE: a cognitive intervention trial to promote independence in older adults. Control Clin Trials. 2001 Aug;22(4):453-79. doi: 10.1016/s0197-2456(01)00139-8. PMID 11514044
- [Background] van Heugten C, Rasquin S, Winkens I, Beusmans G, Verhey F. Checklist for cognitive and emotional consequences following stroke (CLCE-24): development, usability and quality of the self-report version. Clin Neurol Neurosurg. 2007 Apr;109(3):257-62. doi: 10.1016/j.clineuro.2006.10.002. Epub 2006 Nov 28. PMID 17126480
- [Background] Vallat-Azouvi C, Pradat-Diehl P, Azouvi P. The Working Memory Questionnaire: a scale to assess everyday life problems related to deficits of working memory in brain injured patients. Neuropsychol Rehabil. 2012;22(4):634-49. doi: 10.1080/09602011.2012.681110. Epub 2012 Apr 27. PMID 22537095
- [Background] Johnson N, Barion A, Rademaker A, Rehkemper G, Weintraub S. The Activities of Daily Living Questionnaire: a validation study in patients with dementia. Alzheimer Dis Assoc Disord. 2004 Oct-Dec;18(4):223-30. PMID 15592135
- [Background] Wolinsky FD, Vander Weg MW, Howren MB, Jones MP, Dotson MM. A randomized controlled trial of cognitive training using a visual speed of processing intervention in middle aged and older adults. PLoS One. 2013 May 1;8(5):e61624. doi: 10.1371/journal.pone.0061624. Print 2013. PMID 23650501

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention Arm | Control Arm
Started | 20 | 18
Completed | 7 | 7
Not Completed | 13 | 11
Not completed — Never took part in intervention or control arm activities or completed post assessments | 13 | 11

BASELINE CHARACTERISTICS:
Population: 18 subjects in the control arm completed the pre-intervention assessments for CLCE-24, working memory and Activities of daily living.
  20 subjects in the Intervention arm completed the pre-intervention assessments for CLCE-24, and Activities of daily living. 19 subjects completed the working memory assessment.
Groups:
- Intervention Arm: Participants assigned to the intervention/experimental group will undergo twenty training sessions over 10 weeks. In each session, they practice video games selected from Lumosity(http://www.lumosity.com), a web-based cognitive training platform that includes games designed with the purpose of improving the user's cognitive abilities.
- Total: Total of all reporting groups
Arm/Group | Control Arm | Intervention Arm | Total
Number analyzed (Participants) | 18 | 20 | 38
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 16 | 19 | 35
  >=65 years | 2 | 1 | 3
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Data was not collected.
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
CLCE-24 [Mean (Full Range); unit: Number of complaints] — CLCE-24-C, which consists of 13 items (e.g., problems with "doing two things at once" or "remembering new information" . The items involve multiple cognitive domains (including executive functioning, attention, memory, speed of processing and visuospatial perception) and are indicative of the cognitive complaints the patient experiences. The interviewer scores a "0" for the absence of complaints, a "1" for possible complaints and a "2" for the presence of complaints. Total scores range from 0-26 and higher scores indicate more cognitive complaints.
  Number of complaints | 13.7 [8 to 21] | 12.1 [7 to 21] | 12.9 [7 to 21]
Working memory [Mean (Full Range); unit: Units on a Scale] — Working Memory Questionnaire - 30 questions in 3 different domains of 10 questions each. First domain short term storage, second domain was attention, third domain executive aspects of working memory such as decision making, planning ahead or shifting.
  Each question 5 point Likert scale (0-5), three domains, maximal score 50 each for total score out of 150 with higher scores corresponding to more difficulties/complaints. Total score ranges from 0-150, with higher scores corresponding to more difficulties/complaints Population: One subject did not complete the working memory assessment
  Units on a Scale
    number analyzed (Participants) | 18 | 19 | 37
    (all) | 36.17 [8 to 79] | 38 [12.5 to 85] | 37 [8 to 85]
Activity of Daily Living [Mean (Full Range); unit: percentage of impairment] — Activities of daily living: Each answered question was rated on a ﬁve-point Likert-type scale, ranging from 0 (no problem at all) to 4 (very severe problem in everyday life).
  Test is scored by taking the total score of a patient and dividing by the number of items rated and converted to percentiles, allows test to measure deficits seen with regular activities. Total score ranges from 0-100%. Test has a validated cut off points for determine positive results: 0-33% may indicate some impairment, 34-66% moderate impairment, 67+%: severe impairment. Higher values = worse outcomes
  percentage of impairment | 32 [6 to 82] | 23 [6.6 to 55.5] | 27.5 [6 to 82]

OUTCOME MEASURES:

1. Primary Outcome: CLCE-24
Description: Cognitive and Emotional Consequences CLCE-24-C, which consists of 13 items (e.g., problems with "doing two things at once" or "remembering new information" . The items involve multiple cognitive domains (including executive functioning, attention, memory, speed of processing and visuospatial perception) and are indicative of the cognitive complaints the patient experiences. The interviewer scores a "0" for the absence of complaints, a "1" for possible complaints and a "2" for the presence of complaints. Total scores range from 0-26 and higher scores indicate more cognitive complaints.
Time Frame: One year
Population: only 7 subjects in the control arm and 7 subject in the intervention arm participated in the games and completed their post assessment.
Measure: Mean (Full Range); unit: score on scale
Groups:
- Control Arm: Crossword
- Intervention Arm: Lumosity
Arm/Group | Control Arm | Intervention Arm
Number analyzed (Participants) | 7 | 7
score on scale | 12.6 [9 to 14] | 10.4 [7 to 15]

2. Primary Outcome: Working Memory
Description: Working Memory Questionnaire - 30 questions in 3 different domains of 10 questions each. First domain short term storage, second domain was attention, third domain executive aspects of working memory such as decision making, planning ahead or shifting.
  Each question 6 point Likert scale (0-5), three domains, maximal score 50 each for total score out of 150 with higher scores corresponding to more difficulties/complaints. Total score ranges from 0-150, with higher scores corresponding to more difficulties/complaints.
Time Frame: One Year
Population: as for outcome 1
Measure: Mean (Full Range); unit: Units on a scale
Arm/Group | Control Arm | Intervention Arm
Number analyzed (Participants) | 7 | 7
Units on a scale | 35.8 [14 to 51.6] | 31.4 [9.2 to 53.3]

3. Primary Outcome: Activity of Daily Living
Description: Activities of daily living: Each answered question was rated on a ﬁve-point Likert-type scale, ranging from 0 (no problem at all) to 4 (very severe problem in everyday life).
  Test is scored by taking the total score of a patient and dividing by the number of items rated and converted to percentiles, allows test to measure deficits seen with regular activities. Total score ranges from 0-100%. Test has a validated cut off points for determine positive results: 0-33% may indicate some impairment, 34-66% moderate impairment, 67+%: severe impairment. Higher values = worse outcomes
Time Frame: One year
Population: as for outcome 1
Measure: Mean (Full Range); unit: percentage of impairment
Arm/Group | Control Arm | Intervention Arm
Number analyzed (Participants) | 7 | 7
percentage of impairment | 23.7 [10.7 to 35.7] | 18.9 [2.6 to 29.6]

ADVERSE EVENTS:
Time Frame: All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed.
Description: All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed.
Arm/Group | Intervention Arm | Control Arm
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
No subjects analyzed due to incomplete data, leading to unreliable or uninterpretable data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-06-24): https://cdn.clinicaltrials.gov/large-docs/40/NCT02864940/Prot_SAP_000.pdf